CLINICAL TRIAL: NCT01429415
Title: Magnesium Nebulization Utilization in Management of Pediatric Asthma
Acronym: MAGNUMPA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Alberta Children's Hospital (Other); St. Justine's Hospital (Other); Children's Hospital of Eastern Ontario (Other); Stollery Children's Hospital (Other); The Children's Hospital of Winnipeg (Other); Provincial Health Services Authority British Columbia (Other)
Responsible Party: Principal Investigator, Suzanne Schuh, Staff Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1000024908
Record Dates: First submitted 2011-09-02; First posted 2011-09-07 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Acute Asthma
Keywords: pediatric; Acute Asthma; Inhaled Magnesium
MeSH Terms: interventions — Magnesium Sulfate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Group (Experimental): Magnesium Sulfate Sandoz/PPC 600mg and Salbutamol (GlaxoSmithKline/Pharmascience) 5mg by inhalation via Aeroneb Go nebulizer (Philips) with Idehaler Pocket chamber DTF q 20 minutes, 3 treatments.
  Interventions: Drug: Magnesium Sulfate Sandoz
- Control Group (Placebo Comparator): Sodium Chloride USP PPC/Omega (5.5%) placebo and salbutamol GlaxoSmithKline/Pharmascience 5 mg by inhalation via Aeroneb Go nebulizer Philips with Idehaler Pocket chamber DTF q 20 minutes, 3 treatments.
  Interventions: Drug: Sodium Chloride , USP PPC

INTERVENTIONS:
Drug: Magnesium Sulfate Sandoz — Each treatment will utilize 600 mg (1.2 mL) of Magnesium Sulfate Sandoz
  Other Names: Magnesium Sulfate, USP 50% PPC
  Arms: Experimental Group
Drug: Sodium Chloride , USP PPC — Intervention: The control group will receive Sodium Chloride , USP PPC (1.2 mL hypertonic 5.5% saline with 5 mg Salbutamol - GlaxoSmithKline/Pharmascience
  Other Names: Sodium Chloride for Injection USP Omega Laboratories Ltd.
  Arms: Control Group

SUMMARY:
Acute asthma is the most common cause of pediatric hospitalizations. While the investigators know that repeat inhalations of ß2 agonists and ipratropium with early oral steroids substantially reduce hospitalizations, many children are resistant to this standard initial therapy. About a third of children remaining in moderate to severe distress after standard therapy are admitted to hospital and comprise 84% of pediatric acute asthma hospitalizations. Finding safe, non-invasive, and effective strategies to treat children resistant to standard therapy would substantially decrease hospitalizations resulting in considerable health care savings and reduction of the psycho-social burden of the disease. While studies of magnesium sulfate (Mg) given intravenously (IV) suggest that this agent can reduce hospitalizations in both adults and children resistant to standard initial therapy Nebulization is an alternate route for administering Mg. This route has the advantage of being non-invasive and is likely much safer due to lower systemic delivery. Direct delivery via nebulization allows higher Mg concentrations at the target site, the lower airways, with a smaller total drug dose. The investigators propose to conduct a properly designed study to clarify the role of nebulized Mg.

DETAILED DESCRIPTION:
The investigators plan the following specific aims:

1. Primary Objective: To examine if in children with acute asthma remaining in moderate to severe respiratory distress despite maximized initial bronchodilator and steroid therapy there is a reduction in hospitalization rate from the ED in those who receive nebulized Mg with salbutamol versus those receiving salbutamol only.

   Hypothesis: The investigators hypothesize that the children with Pediatric Respiratory Assessment Measure (PRAM) ≥ 5 points after optimized initial inhaled bronchodilator and oral steroid therapies who are given nebulized Mg in addition to nebulized salbutamol will have significantly lower hospitalization rate within 24 hours of starting the study compared to those given salbutamol only.
2. To compare a difference in the changes in the validated Pediatric Respiratory Assessment Measure (PRAM), respiratory rate, oxygen saturation and blood pressure from randomization baseline to 240 minutes in the two groups
3. To determine if there is a significant association between the difference in the primary outcome between the groups and the patient's age, gender, baseline PRAM score, personal history of atopy and "viral-induced wheeze" phenotype.

Hypothesis(es) to be Tested In this randomized, double-blind seven-centre trial, the investigators hypothesize that children with acute asthma with a Pediatric Respiratory Assessment Measure (PRAM) of ≥ 5 points after optimized initial inhaled bronchodilator and oral steroid therapies who are given nebulized Mg in addition to nebulized salbutamol will have at least a 10% lower hospitalization rate within 24 hours of starting the study as compared to those given salbutamol only.

ELIGIBILITY:
Inclusion Criteria:

1. 2-17 years of age
2. Diagnosis of asthma/reactive airways/viral wheeze, defined as this diagnosis made by a physician and at least one prior acute episode of wheezing with cough or dyspnea treated with inhaled ß2 agonists or oral corticosteroids. Our study population will exclude bronchiolitis and first-time wheeze (potential alternate diagnoses).
3. Persistent moderate to severe airway obstruction after 3 doses of salbutamol and ipratropium (as per site specific standard of care guidelines) -, defined as a PRAM 5 or higher. A PRAM score of 5 or more following initial therapy indicates the child has at least moderate disease severity and has a high likelihood of being hospitalized.This group of children includes 84% of all pediatric asthma hospitalizations; therefore, finding an effective therapy for this population has great potential to significantly reduce hospitalizations. (Appendix B).

Exclusion Criteria:

1. No previous history of wheezing or bronchodilator therapy. Some children who present with wheezing for the first time will have other diagnoses which would not be expected to respond to Mg.
2. Patients who have already received IV Mg therapy during the index visit.
3. Critically ill children requiring immediate intubation. These children need immediate ICU management and hospitalization.
4. Children who in the opinion of the treating physician require a chest radiograph due to atypical clinical presentation and are found to have radiologist-confirmed pneumonia. These rare patients may have to be hospitalized primarily for treatment of the infection and may not respond to magnesium.
5. Known co-existent renal, chronic pulmonary, neurologic, cardiac or systemic disease. These conditions may influence the response to Mg and hospitalization.
6. Known hypersensitivity to Mg sulfate.
7. Patients previously enrolled in the study.
8. Insufficient command of the English and or French language.
9. Lack of a home or cellular telephone.
10. Known allergy/sensitivity to latex.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 818 (Actual)
Dates: Start 2011-09-26 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
Hospitalization of Subject | Up to 24 hours after treatment
  Defined as admission to an inpatient unit within 24hours of the start of experimental therapy due to continued/worsening distress.

SECONDARY OUTCOMES:
Pediatric Respiratory Assessment Measure (PRAM) | 0, 20, 40 60, 120, 180, 240 minutes post dose
  PRAM is a validated measure of asthma severity in the Emergency Department
Changes in Vitals | 0, 20, 40, 60, 120, 180, 240 minutes post dose
  Respiratory Rate, O2 saturation, Blood pressure
Number of Salbutamol Treatments | Up to 240 minutes post dose
  This measure of additional therapy may strengthen the measure of benefit of inhaled magnesium
Medical History and Phenotype | Baseline
  The investigators will measure hospitalization and age, gender, pre-randomization PRAM score, personal history of atopy, and "acute viral induced wheeze" phenotype. This phenotype will be defined by age less than 5 years, co-existent upper respiratory tract infection, no interval symptoms between exacerbations, no atopy

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Schuh, MD, Principal Investigator — The Hospital for Sick Children
Locations (7):
- Canada (7):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Hospital, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - The Manitoba Institute of Child Health, Winnipeg, Manitoba
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Ste Justine Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schuh S, Freedman SB, Zemek R, Plint AC, Johnson DW, Ducharme F, Gravel J, Thompson G, Curtis S, Stephens D, Coates AL, Black KJ, Beer D, Sweeney J, Rumantir M, Finkelstein Y; Pediatric Emergency Research Canada. Association Between Intravenous Magnesium Therapy in the Emergency Department and Subsequent Hospitalization Among Pediatric Patients With Refractory Acute Asthma: Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2021 Jul 1;4(7):e2117542. doi: 10.1001/jamanetworkopen.2021.17542. PMID 34279646
- [Derived] Schuh S, Sweeney J, Rumantir M, Coates AL, Willan AR, Stephens D, Atenafu EG, Finkelstein Y, Thompson G, Zemek R, Plint AC, Gravel J, Ducharme FM, Johnson DW, Black K, Curtis S, Beer D, Klassen TP, Nicksy D, Freedman SB; Pediatric Emergency Research Canada (PERC) Network. Effect of Nebulized Magnesium vs Placebo Added to Albuterol on Hospitalization Among Children With Refractory Acute Asthma Treated in the Emergency Department: A Randomized Clinical Trial. JAMA. 2020 Nov 24;324(20):2038-2047. doi: 10.1001/jama.2020.19839. PMID 33231663
- [Derived] Schuh S, Sweeney J, Freedman SB, Coates AL, Johnson DW, Thompson G, Gravel J, Ducharme FM, Zemek R, Plint AC, Beer D, Klassen T, Curtis S, Black K, Nicksy D, Willan AR; Pediatric Emergency Research Canada Group. Magnesium nebulization utilization in management of pediatric asthma (MagNUM PA) trial: study protocol for a randomized controlled trial. Trials. 2016 May 24;17(1):261. doi: 10.1186/s13063-015-1151-x. PMID 27220675